CLINICAL TRIAL: NCT06083181
Title: A Multicenter, Prospective, Open-label Clinical Trial to Evaluate the Safety and Effectiveness of the Perf-Fix Otologic Gel Patch to Aid in the Repair of Chronic Tympanic Membrane Perforation
Brief Title: Perf-Fix Study for Chronic Tympanic Membrane Repair
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tympanogen (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYMP001; 2SB1DC018255-02 (NIH); 1203 (Other Grant/Funding Number: VA Catalyst)
Record Dates: First submitted 2023-09-11; First posted 2023-10-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Tympanic Membrane Perforation
Keywords: tympanic membrane; eardrum; pediatric; tympanoplasty; myringoplasty
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment group (Experimental): Treatment group receives one application of Perf-Fix
  Interventions: Device: Perf-Fix Otologic Gel Patch

INTERVENTIONS:
Device: Perf-Fix Otologic Gel Patch — Gel patch application
  Other Names: Perf-Fix

SUMMARY:
The purpose of the study is to assess the effectiveness of Perf-Fix as a gel patch to aid in the natural healing process to close chronic, >25% tympanic membrane perforation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent, legally authorized representative (LAR) consent, or LAR consent and assent when age appropriate
* Females and males at least 5 years old
* Perforation involves >25% of the tympanic membrane
* Perforation has not spontaneously closed after 4 weeks of watchful waiting
* Perforation is not actively healing
* Perforation can be visualized by an endoscope or microscope
* Ear wax does not occlude the perforation

Exclusion Criteria:

* Perforation is marginal (a perforation that has an area with no tympanic membrane between the perforation and the bony canal)
* Active otitis media, with or without effusion
* Otorrhea from the middle ear for more than 3 months
* History of cleft palate
* Receiving radiation therapy or taking corticosteroids, immunosuppressive agents, or chemotherapy
* Currently taking systemic antibiotics, antibiotic ear drops, and/or steroid ear drops
* Current bacterial or viral infection
* Fever (Temperature >100°F) at time of index procedure
* Diagnosed with cholesteatoma mass in the tympanic cavity
* Known history of malignant ear canal tumors within 3 years of screening for eligibility
* Abrasions/lacerations to the external auditory canal
* Significant medical condition that could prevent full participation in the procedures required for the study
* Investigator feels the subject will be unable to cooperate with the application procedure
* Parent/LAR feels the subject will be unable to cooperate with the application procedure
* Allergy to shellfish
* Known to be or could be pregnant
* Adults lacking capacity to consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Eardrum closure | 12 weeks
  The rate of success in Perf-Fix closing perforated eardrums. Success is defined as closure of the perforation.
Device- and procedure-related safety | 12 weeks
  Incidence of adverse events over the course of the study for each subject.

SECONDARY OUTCOMES:
Procedural success | 1 hour
  Perf-Fix is successfully applied by the clinician to the subject's eardrum perforation, measured as Yes/No.
  Procedural Success (ALL steps accomplished):
  * complete device preparation
  * apply device to tympanic membrane perforation
  * complete curing process using light guide and curing light
  * visualize cured device on tympanic membrane perforation
  * subject recovers from procedure
  Procedural Failure (including but not limited to):
  * inability to apply device to tympanic membrane perforation
  * device does not adhere to tympanic membrane
  * behavioral intolerance to procedure
  * all steps for Procedural Success not completed
Perforation size - percent area | 1 hour
  Size of perforation measured in percent area of eardrum.
Perforation size - length and width | 1 hour
  Size of perforation measured in mm across length and width of perforation.
Perforation location | 12 weeks
  Quadrant(s) of perforation location: Anterosuperior, anteroinferior, posterosuperio, and/or posteroinferior
Time of procedure | 1 hour
  Time taken to apply Perf-Fix in single application
Time to heal | 12 weeks
  Time from Perf-Fix application to tympanic membrane healing
Air-bone gap | 12 weeks
  Measurement of air-bone gap by audiogram at 500, 1000, and 2000 Hz
Word recognition | 12 weeks
  Measurement of hearing ability by percent of words correctly recognized
Tympanometry | 12 weeks
  Measurement of tympanic membrane integrity as normal or abnormal
Procedure tolerability | 1 hour
  Assess pain/discomfort using Visual Analogue Scale before and after each Perf-Fix application procedure on a scale 0-10 (0=no pain, 10=unbearable pain)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - House Institute, Los Angeles, California
  - Advanced ENT & Allergy, Louisville, Kentucky
  - South Louisiana Ear, Nose, and Throat, Mandeville, Louisiana
  - Mass Eye and Ear, Boston, Massachusetts
  - Carolina Ear & Hearing Clinic, Raleigh, North Carolina
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No